CLINICAL TRIAL: NCT05773716
Title: The Effects of Combination Therapy With Electroacupuncture and Pelvic Floor Muscle Training on Stress Urinary Incontinence Following Radical Prostatectomy: A Randomized Controlled Trial
Brief Title: Electroacupuncture and Pelvic Floor Muscle Training for Male Stress Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RenJi Hospital (Other)
Collaborators: Longhua Hospital (Other)
Responsible Party: Principal Investigator, Qi-Xiang Song, Principal Investigator, RenJi Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ST2023
Record Dates: First submitted 2023-01-19; First posted 2023-03-17 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Stress Urinary Incontinence
Keywords: Incontinence; Radical prostatectomy; Men; Pelvic floor muscle training; Acupuncture; Bladder diary; Pad test
MeSH Terms: conditions — Urinary Incontinence, Stress; Multiple Endocrine Neoplasia Type 1 | interventions — Electroacupuncture

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Electroacupuncture plus pelvic floor muscle training (Experimental): Participants in this arm will receive pelvic floor muscle training using unified standards, and electroacupuncture therapy for 6 weeks.
  Interventions: Behavioral: Pelvic floor muscle training; Other: Electroacupuncture
- Sham electroacupuncture plus pelvic floor muscle training (Sham Comparator): Participants in this arm will receive pelvic floor muscle training using the same approach as that in experimental group, and sham electroacupuncture for 6 weeks.
  Interventions: Behavioral: Pelvic floor muscle training; Other: Sham electroacupuncture

INTERVENTIONS:
Behavioral: Pelvic floor muscle training — Participants will receive daily pelvic floor muscle training for 6 consecutive weeks. In specific, they will be instructed to perform 3 training sessions (morning, afternoon and evening) per day with an emptied bladder in a relaxed state. During each session, 10 muscle stretches are required with each contraction duration of 2~6-second and a 2~6-second relaxation following each one.
Other: Electroacupuncture — Participants will also receive electroacupuncture at bilateral Zhongliao (BL33), Huiyang (BL35), Zhongji (CV3), Guanyuan (CV4) and Dahe (KI12). During each therapy session, the electroacupuncture stimulation of acupoints in the abdomen and sacral regions will last for 30 minutes in total (15 minutes for each region) with a continuous wave of 50 Hz and a current intensity of 1 to 5 mA (preferably with the skin around the acupoints shivering mildly without pain). Participants will receive 3 treatment sessions per week (ideally every other day) for 6 consecutive weeks, 18 sessions in total.
  Arms: Electroacupuncture plus pelvic floor muscle training
Other: Sham electroacupuncture — Sham electroacupuncture will be carried out with pragmatic placebo needles on the same acupoints in the experimental group. Procedures, electrode placements, and other treatment settings will also stay the same but with no electrical stimulation output.
  Arms: Sham electroacupuncture plus pelvic floor muscle training

SUMMARY:
The goal of this clinical study is to compare the effects of combined electroacupuncture with pelvic floor muscle training (PFMT) versus PFMT alone in the treatment of involuntary urine leakage following prostate removal procedure due to prostate cancer. The main goal is to determine that whether adding electroacupuncture to PFMT provides extra benefits in relieving urinary leakage and improves patients' quality of life. All participants will be required to perform daily PFMT for 6 weeks using uniformed standards. During the meantime, those assigned to the experimental group will additionally receive electroacupuncture three times per week for 6 weeks, while those in control group will receive sham treatment with same duration. Researchers will compare the urine leakage severity between the two groups to see if adding electroacupuncture can facilitate the recovery of symptom.

DETAILED DESCRIPTION:
This randomized controlled trial will recruit patients presenting stress urinary incontinence 6 weeks after radical prostatectomy, with the aim to determine whether adding electroacupuncture therapy to pelvic floor muscle training (PFMT) provides extra benefits in relieving stress urinary incontinence following radical prostatectomy. Followed by signing the informed consent and baseline assessments, participants with be randomly allocated to either PFMT plus electroacupuncture arm or PFMT plus sham electroacupuncture arm in a 1:1 ratio.

Pelvic floor muscle training will be conducted daily using a consistent approach. In short, before training, the patients are required to empty the bladder and relax the whole body in a sitting or lying position. The contraction of the pelvic floor muscles is maintained for 2-6 seconds, followed by a relaxation for 2-6 seconds. This process is repeated 10 times per session, three sessions per day (in the morning, afternoon and evening), and performed daily for 6 continuous weeks.

Electroacupuncture will be performed at bilateral Zhongliao, Huiyang, Zhongji, Guanyuan and Dahe, three treatment sessions per week for 6 consecutive weeks. For sham electroacupuncture, The same acupoints will be punctured as that in treatment group, except the use of blunt-tipped needles (identical in appearance compared with normal needles) to puncture through the fixed pad and to reach the skin surface. In both groups, the needles will be clamped by electrodes which are connected to a pulse generator (Huatuo SDZ- EA, Suzhou, China). In consistency with our previous settings, continuous wave with frequency of 50Hz will be used. The current intensity is gradually increased ranging from 1mA to 5mA, according to the patient's tolerance.

Patients will be appraised at baseline, 3, 6, 10 and 18 weeks after the initiation of treatments to determine the changes of incontinence symptom, quality of life and pelvic structures. The primary outcome is the change of urine leakage amount during a 1-hour pad test at 6-week timepoint. The secondary outcomes include parameters derived from the International Consultation on Incontinence Modular Questionnaire - urinary incontinence short form, mean 24-hour pad use, pelvic magnetic resonance imaging (except for those with contraindications, such as metallic implants or psychological disorders), and the documentation of adverse events.

The statistical analysis of the baseline and outcomes at each timepoint is based on the intention-to-treat population. In addition, the data analysis of the primary outcome is also based on the per-protocol population as a supportive analysis. Quantitative variables will be compared using either independent t-tests or Mann-Whitney U-tests based on their normality. The statistical significance between nominal variables will be detected using Pearson's chi-squared tests or Fisher's exact tests. Statistical analysis will be performed using both SPSS software and R package, and the level of significance will be set at <0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients present stress urinary incontinence 6 weeks after radical prostatectomy
* Aged between 45-80 years
* With an urine leakage amount over 1g measured by the one-hour pad test
* Participate voluntarily with signed the informed consent

Exclusion Criteria:

* The existence of stress urinary incontinence symptoms before the surgery
* Urine leakage due to urgency incontinence, voiding dysfunction, nocturnal enuresis and fistula
* Known history of radiation therapy to the pelvic region
* Evidence of tumor recurrence or metastasis
* Those who have already underwent treatment for stress urinary incontinence
* Patients with hemorrhagic disease or hemorrhagic tendency
* The presence of ulcer, abscess and skin infection at locations of target acupoints
* With histories of cardiac pacemaker, intravascular stent and metal allergy
* With poor health conditions due to coexisting of acute comorbidities of the heart, brain, lung and kidney
* Those who refuse to sign the informed consent and unable to comply with the study protocol

Ages: 45 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
The change of urine leakage amount at 6 weeks | measured at baseline and 6 weeks after treatment
  The 1-hour pad test will be applied to quantitatively measure the changes of the urine leakage severity. In specific, patients will be asked to wear pre-weighed pads and drink 500 ml of sodium-free liquid in <15 minutes. After rest, they are instructed to exercise for 30 minutes, including: walking, climbing up and down one ﬂight of stairs, standing-up from sitting (10 times), coughing vigorously (10 times), running on the spot for 1 minute, bending to pick up an object from the ﬂoor (5 times) and washing hands for 1 minute in running water. Before and after the test, the weight of the pad is measured with a high-precision balance in order to determine the amount of leakage. For this test, an increase of 1 to 10 g represents mild incontinence, 11 to 50 g represents moderate incontinence, and >50 g represents severe incontinence.

SECONDARY OUTCOMES:
One-hour pad test at 3, 10, 18 weeks | measured at 3, 10 and 18 weeks after treatment
  For the 1-hour pad test, patients will be asked to wear pre-weighed pads and drink 500 ml of sodium-free liquid in <15 minutes. After rest, they are instructed to exercise for 30 minutes, including: walking, climbing up and down one ﬂight of stairs, standing-up from sitting (10 times), coughing vigorously (10 times), running on the spot for 1 minute, bending to pick up an object from the ﬂoor (5 times) and washing hands for 1 minute in running water. Before and after the test, the weight of the pad is measured with a high-precision balance in order to determine the amount of leakage. For this test, an increase of 1 to 10 g represents mild incontinence, 11 to 50 g represents moderate incontinence, and >50 g represents severe incontinence.
The status of 24-hour pad use | measured at baseline, 6 and 18 weeks after treatment
  The 24-hour pad use will be recorded as the average daily pad number in three continuous days
Urinary incontinence questionnaires | measured at baseline, 3, 6, 10 and 18 weeks after treatment
  The patient-reported continence status will be evaluated by the International Consultation on Incontinence Modular Questionnaire - urinary incontinence short form (ICIQ-UI-SF). The total score will be calculated based on three questions, namely the frequency of leakage (scores from 0 to 5 points), the amount of leakage (scores 0, 2, 4 or 6 points) and the impact of leakage (scores from 0 to 10 points).
Pelvic Magnetic resonance imaging | measured at baseline, 6 and 18 (optional) weeks after treatment
  The pelvic magnetic resonance imaging (MRI) will be performed with a 1.5-T scanner with the patients in a supine position. The imaging protocol included a transversal T1-weighted 2D gradient echo sequence. High-spatial-resolution T2-weighted TSE sequences will be obtained in the axial, coronal and sagittal orientation. Several parameters will be measured, including membranous urethral length (mm), urethral wall thickness (mm), levator ani muscle thickness (mm), obturator internus muscle thickness (mm) etc. Besides, the position of the bladder neck, the shape of the bladder and the presence of a dilated posterior urethra will also be recorded. The MRI can be waived if contraindications are noted, such as metallic implants or psychological disorders.
Adverse events | measured at 3, 6, 10 and 18 weeks after treatment
  Although electroacupuncture is well-known as a minimally invasive therapy which can be carried out in the clinic, the adverse events will be carefully documented by the researchers base on the patients' subjective report.
Data of birth | documented at baseline
  The date of birth will be recorded as year/month/date.
Height | documented at baseline
  The height will be measured in meters.
Weight | documented at baseline
  The weight will be measured in kilograms.
Body mass index (BMI) | documented at baseline
  The BMI is calculated as weight (kg) / height (m^2)
Comorbidites | documented at baseline
  The comorbidities, such as hypertension, diabetes and stroke etc., will be recorded by patient-self report.
The duration after radical prostatectomy | documented at baseline
  The duration is calculated as the days between the date of recruitment and the date of radical prostatectomy.
The TNM tumor staging | documented at baseline
  The TNM tumor staging is recorded according to the pathology report after radical prostatectomy.
The radical prostatectomy technique | documented at baseline
  Whether the neurovasulcar preservation technique and lymph node dissection was performed is achieved according to the surgery record.
The presence of positive surgical margin | documented at baseline
  This is recorded according to the pathology report after radical prostatectomy.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Xue, MD, Study Chair — Department of Urology, Ren Ji Hospital, Shanghai Jiao Tong University School of Medicine; Yuelai Chen, MD, Study Chair — Shanghai University of Traditional Chinese Medicine
Locations (1):
- Renji Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
The IPD will be made available to other researchers upon reasonable request after the publication of this trial.
Supporting Information: Study Protocol
Time Frame: The study protocol will be ready to share upon reasonable request after the publication of study.

REFERENCES:
- [Background] Tang K, Su T, Fu L, Chen Z, Liu G, Hou W, Ming S, Song Q, Feng S, Liu X, Wang R, Liu B, Chen Y. Effect of Electroacupuncture Added to Pelvic Floor Muscle Training in Women with Stress Urinary Incontinence: A Randomized Clinical Trial. Eur Urol Focus. 2023 Mar;9(2):352-360. doi: 10.1016/j.euf.2022.10.005. Epub 2022 Oct 26. PMID 36420937
- [Background] Liu Z, Liu Y, Xu H, He L, Chen Y, Fu L, Li N, Lu Y, Su T, Sun J, Wang J, Yue Z, Zhang W, Zhao J, Zhou Z, Wu J, Zhou K, Ai Y, Zhou J, Pang R, Wang Y, Qin Z, Yan S, Li H, Luo L, Liu B. Effect of Electroacupuncture on Urinary Leakage Among Women With Stress Urinary Incontinence: A Randomized Clinical Trial. JAMA. 2017 Jun 27;317(24):2493-2501. doi: 10.1001/jama.2017.7220. PMID 28655016
- [Background] Su T, Zhou J, Liu Z, Chen Y, Zhang W, Chu H, Luo Q, Lu J, An J, Liu B. The efficacy of electroacupuncture for the treatment of simple female stress urinary incontinence - comparison with pelvic floor muscle training: study protocol for a multicenter randomized controlled trial. Trials. 2015 Feb 8;16:45. doi: 10.1186/s13063-015-0560-1. PMID 25887231
- [Background] Geraerts I, Van Poppel H, Devoogdt N, Joniau S, Van Cleynenbreugel B, De Groef A, Van Kampen M. Influence of preoperative and postoperative pelvic floor muscle training (PFMT) compared with postoperative PFMT on urinary incontinence after radical prostatectomy: a randomized controlled trial. Eur Urol. 2013 Nov;64(5):766-72. doi: 10.1016/j.eururo.2013.01.013. Epub 2013 Jan 21. PMID 23357349
- [Background] Ribeiro LH, Prota C, Gomes CM, de Bessa J Jr, Boldarine MP, Dall'Oglio MF, Bruschini H, Srougi M. Long-term effect of early postoperative pelvic floor biofeedback on continence in men undergoing radical prostatectomy: a prospective, randomized, controlled trial. J Urol. 2010 Sep;184(3):1034-9. doi: 10.1016/j.juro.2010.05.040. PMID 20643454
- [Derived] Bi X, Chen Y, Wu R, Gao W, Fan Q, Wang S, Pan J, Xue W, Song QX, Tang K. The effects of combination therapy with electroacupuncture and pelvic floor muscle exercise on stress urinary incontinence following radical prostatectomy: the protocol for a randomized controlled trial. Front Surg. 2025 Dec 16;12:1490210. doi: 10.3389/fsurg.2025.1490210. eCollection 2025. PMID 41477477